CLINICAL TRIAL: NCT00231660
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study of the Efficacy and Safety of Topiramate in the Treatment of Obese, Type 2 Diabetic Patients Treated With Metformin
Brief Title: A Study of the Efficacy and Safety of Topiramate in the Treatment fo Obese, Type 2 Diabetic Patients Treated With Metformin
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR003718
Record Dates: First submitted 2005-09-30; First posted 2005-10-04 (Estimated); Last update posted 2011-06-08 (Estimated); Status verified 2011-01

CONDITIONS: Obesity; Diabetes Mellitus, Type 2; Diabetes Mellitus, Adult-Onset
Keywords: Type 2 Diabetes; Obesity; Metformin; Hemoglobin A1c; Adult-Onset Diabetes Mellitus (AODM)
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2 | interventions — Topiramate

INTERVENTIONS:
Drug: topiramate

SUMMARY:
The purpose of this study is to compare the efficacy (in terms of weight and hemoglobin type A1c [HbA1c]) and safety of topiramate (96 milligrams[mg] or 192 mg daily) with placebo in the treatment of obesity in Type 2 diabetic patients receiving metformin.

DETAILED DESCRIPTION:
Topiramate is not approved for the treatment of obesity. This double-blind, placebo-controlled study is designed to assess the efficacy and safety of topiramate in Type 2 diabetic patients with obesity who are well-controlled on metformin alone. Patients are randomized to receive either topiramate (up to a target dose of 96 or 192 mg per day) or placebo for one year. Assessments of efficacy include weight reduction, levels of HbA1c (shows average blood sugar level over a few months), Body Mass Index (BMI), and Health Related Quality of Life (HRQOL) measures. Safety evaluations (incidence of adverse events, vital signs, hypoglycemic events, electrocardiograms [ECGs], clinical laboratory values) are monitored throughout the study. The study hypothesis is that topiramate, combined with metformin and non-pharmacologic therapy, can effectively achieve significant weight reduction and is well tolerated. During the first 8 weeks, oral doses of matching placebo or topiramate are increased gradually to target dose (96 milligrams[mg] or 192mg daily); the dose will be maintained for 1 year, then gradually reduced and stopped

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Type 2 diabetes and receiving metformin monotherapy for at least the previous 4 months and on a stable daily dose for at least 2 months prior to enrollment
* Metformin total daily dose not to exceed 2.1 grams/day
* Body Mass Index >= 27 and < 50
* HbA1c < 11%
* Fasting plasma glucose >= 126 and < 240
* Stable weight
* Female patients must be postmenopausal for at least 1 year, surgically incapable of childbearing, or practicing an acceptable method of contraception (requires negative pregnancy test)

Exclusion Criteria:

* Known contraindication, or hypersensitivity to topiramate
* Use of other antidiabetic medications within the last 4 months
* Excessive weight loss
* Diagnosis of type 1 diabetes
* History of severe or recurrent hypoglycemic episodes
* Severe pulmonary disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 211 (Actual)
Dates: Start 2000-10; Study Completion 2002-06 (Actual)

PRIMARY OUTCOMES:
The percent change in body weight and change in HbA1c from baseline (Week 0) to one year after maintenance therapy (Week 60).

SECONDARY OUTCOMES:
Changes from baseline or from enrollment to Week 60 in BMI and HRQOL measures; safety evaluations, such as adverse events and vital signs throughout study.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- See also: A Study of the Efficacy and Safety of Topiramate in the Treatment of Obese, Type 2 Diabetic Patients Treated with Metformin — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=538&filename=CR003718_CSR.pdf